CLINICAL TRIAL: NCT02035293
Title: Frequency of Diagnostic Symptomatic Pulmonary Embolism's in Patients Hospitalized for Clinical Exacerbation of Chronic Obstructive Pulmonary Disease (COPD)
Acronym: PEP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PEP; RB 13-087 [CHRU Brest]
Record Dates: First submitted 2014-01-03; First posted 2014-01-14 (Estimated); Last update posted 2025-12-03 (Actual); Status verified 2017-12

CONDITIONS: Chronic Obstructive Pulmonary Disease; Patients Hospitalized for a COPD Exacerbation
Keywords: COPD Exacerbation; Pulmonary embolism; Standardized and consensus diagnostic strategy
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Pulmonary Embolism

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- PEP (Other): No drug and no placebo were used in this study. For all the patients who participated at the study PEP, only following exams must be performed: a clinical probability score (revised Geneva score), plasma D-dimer assay and if necessary, a chest multidetector-row CT angiography and venous ultrasound of the lower limbs
  Interventions: Other: PEP

INTERVENTIONS:
Other: PEP
  Other Names: No drug and no placebo were used in this study. For all the patients who participated at the study PEP, only exams must be performed;

SUMMARY:
A standardized diagnostic strategy of pulmonary embolism will be applied to eligible patients, incorporating a clinical probability score (revised Geneva score), plasma D-dimer assay and if necessary, a multidetector-row CT angiography thoracic and venous ultrasound of the lower limbs. All the patient with a pulmonary embolism diagnosed or not, will be followed for 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients hospitalized for a COPD exacerbation
* COPD previously diagnosed

Exclusion Criteria:

* Allergy to iodinated contrast
* Creatinine clearance < 30 mL / min
* Patient hospitalized for exacerbation of COPD for more than 48 hours
* Pneumothorax
* Exams impossible to be performed
* Pregnancy
* Life expectancy < 3 months
* Patients already receiving anticoagulant therapy for another reason (mechanical valve, cardiac arrhythmia).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 750 (Actual)
Dates: Start 2014-01-08 (Actual); Primary Completion 2017-10-13 (Actual); Study Completion 2017-10-13 (Actual)

PRIMARY OUTCOMES:
Frequency of pulmonary embolism in patients hospitalized for a clinical exacerbation of COPD. | 27 months

SECONDARY OUTCOMES:
The rate of pulmonary embolism diagnosed during the 3 month follow-up in patients whom pulmonary embolism was initially excluded when they've been included in the study | 27 months

CONTACTS AND LOCATIONS:
Overall Officials: Francis COUTURAUD, PU-PH, Principal Investigator — CHRU de Brest
Locations (7):
- France (7):
  - CHU, Angers
  - CHRU de Brest, Brest
  - HIA, Brest
  - CHU Clermont-Ferrand, Clermont-Ferrand
  - Hôpital Européen Georges Pompidou, Paris
  - CH de Cornouaille Quimper, Quimper
  - Hôpital Nord, Saint-Etienne

REFERENCES:
- [Result] Couturaud F, Bertoletti L, Pastre J, Roy PM, Le Mao R, Gagnadoux F, Paleiron N, Schmidt J, Sanchez O, De Magalhaes E, Kamara M, Hoffmann C, Bressollette L, Nonent M, Tromeur C, Salaun PY, Barillot S, Gatineau F, Mismetti P, Girard P, Lacut K, Lemarie CA, Meyer G, Leroyer C; PEP Investigators. Prevalence of Pulmonary Embolism Among Patients With COPD Hospitalized With Acutely Worsening Respiratory Symptoms. JAMA. 2021 Jan 5;325(1):59-68. doi: 10.1001/jama.2020.23567. PMID 33399840